CLINICAL TRIAL: NCT01237951
Title: High-dose Gemcitabine, Busulfan and Melphalan With Autologous Hematopoietic-Cell Support for Patients With Poor-Risk Myeloma
Brief Title: High-Dose Gemcitabine, Busulfan and Melphalan With Hematopoietic-Cell Support for Patients With Poor-Risk Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0506; NCI-2012-01906 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Myeloma
Keywords: Autologous Hematopoietic-Cell Support; Stem Cell Transplant; Busulfan; Myleran; Busulfex; Gemcitabine; Gemzar; Melphalan; Alkeran; Decadron; Dexamethasone; G-CSF; Filgrastim; Neupogen
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Fibroblast Growth Factor 7; Dexamethasone; Calcium Dobesilate; Gemcitabine; Busulfan; Melphalan; Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GemBuMel (Experimental): Gemcitabine 1875 mg/m^2 IV (75 mg/ m2 bolus followed by 1800 mg/m^2 over 3 hours) on Day -8 and Day -3 as an outpatient or inpatient.
  Busulfan 32 mg/m2 test dose with PKs as outpatient before Day -12, or as an inpatient on Day -10.
  Busulfan area under curve (AUC) 4,000 by vein on Days -8 to -5 as an outpatient or inpatient.
  Melphalan 60 mg/m^2 IV on Days -3 and -2 over 30 minutes on both days as an outpatient or inpatient.
  Palifermin 60 micrograms/kg infused as an IVP (by vein) over 15-30 seconds Days -12 to -10 and Days 0 to +2 as an outpatient.
  Palifermin 60 micrograms/kg by vein on Days -13 to -11 and on Days 0, +1 and +2 as in inpatient.
  Dexamethasone 8 mg IV twice a day by vein over 15 minutes Days -9 through -2 as an outpatient or inpatient. G-CSF 5 mcg/kg/day subcutaneously beginning on Day +5 and continuing until neutrophil recovery is documented.
  Stem Cell Transplant: On Day 0, stem cells returned to body by vein over 30-60 minutes.
  Interventions: Drug: Palifermin; Drug: Dexamethasone; Drug: Gemcitabine; Drug: Busulfan; Drug: Melphalan; Procedure: Stem Cell Transplant; Drug: G-CSF

INTERVENTIONS:
Drug: Palifermin — 60 micrograms/kg infused as an IVP (by vein) over 15-30 seconds Days -12 to -10 and Days 0 to +2 as an outpatient.
  60 micrograms/kg by vein on Days -13 to -11 and on Days 0, +1 and +2 as in inpatient.
  Other Names: kepivance
Drug: Dexamethasone — 8 mg IV twice a day by vein over 15 minutes Days -9 through -2 as an outpatient or inpatient.
  Other Names: decadron
Drug: Gemcitabine — 1875 mg/m^2 IV (75 mg/ m2 bolus followed by 1800 mg/m^2 over 3 hours) on Day -8 and Day -3 as an outpatient or inpatient.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Busulfan — 32 mg/m2 test dose with PKs as outpatient before Day -12, or as an inpatient on Day -10.
  Busulfan AUC 4,000 by vein on Days -8 to -5 as an outpatient or inpatient.
  Other Names: myleran; busulfex
Drug: Melphalan — 60 mg/m^2 IV on Days -3 and -2 over 30 minutes on both days as an outpatient or inpatient.
  Other Names: Alkeran
Procedure: Stem Cell Transplant — On Day 0, stem cells returned to body by vein over 30-60 minutes.
  Other Names: SCT; ASCT
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning on Day +5 and continuing until neutrophil recovery is documented.
  Other Names: Filgrastim; Neupogen

SUMMARY:
The goal of this clinical research study is to learn if the combination of gemcitabine, busulfan, and melphalan, when given before a stem cell transplant, can help to control refractory myeloma. The safety of this study treatment will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Busulfan and melphalan are designed to bind to the DNA (genetic material) of cells, which may cause cancer cells to die. They are commonly used in stem cell transplantation.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may help to increase the effect of busulfan and melphalan on cancer cells by not allowing these cells to repair the DNA damage caused by busulfan or melphalan.

Busulfan Test Dose:

You will receive a test dose of busulfan by vein over about 60 minutes. This low-level test dose of busulfan is to check how the level of busulfan in your blood levels changes over time. This information will be used to decide the next dose needed to reach the target blood level that matches your body size. You will most likely receive this as an outpatient during the week before you are admitted to the hospital. If it cannot be given as an outpatient, you will be admitted to the hospital on Day -11 (11 days before your stem cells are returned to your body) and the test dose will be given on Day -10.

About 11 samples of blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points and will help the study doctor determine what your dose of busulfan should be on study. These blood samples will be drawn at various timepoints before you receive busulfan and over about the next 11 hours. The blood samples will be repeated again on the first day of high-dose busulfan treatment Day -8. A temporary heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed, you will receive the standard dose of busulfan.

If you receive the busulfan test dose as an outpatient:

On Days -12 (12 days before your stem cells are returned to your body) through Day -10, you will receive palifermin by vein over about 30 seconds to help decrease the risk of side effects in the mouth and throat.

You will be admitted on Day -9 and will receive fluids by vein to hydrate you. You will swish the liquids caphosol and glutamine in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. These drugs are also used to help decrease the risk of side effects in the mouth and throat.

On Days -8 through -5, you will receive busulfan by vein over about 3 hours.

On Days -8 and -3, you will receive gemcitabine by vein over about 3 hours.

On Day -4, you will not receive any drugs.

If you receive the busulfan test dose as an inpatient:

On Days -13 through Day -11, you will receive palifermin by vein over about 30 seconds each day to help decrease the risk of side effects in the mouth and throat.

You will be admitted on Day -11 and will receive fluids by vein to hydrate you. You will swish the liquids caphosol and glutamine in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. These drugs are also used to help decrease the risk of side effects in the mouth and throat.

On Day -10, you will receive the busulfan test dose by vein over 45 minutes.

On Day -9, you will not receive any drugs.

On Days -8 and -3, you will receive gemcitabine by vein over about 3 hours on both days.

On Days -8 through -5, you will receive busulfan by vein over about 3 hours each day.

Study Drug Administration (for all patients):

On Days -9 through -2, you will receive dexamethasone by vein over about 15 minutes to help decrease the risk of the possible side effects of the study drugs.

On Days -3 and -2, you will receive melphalan by vein over about 30 minutes on both days.

On Day -1, you will not receive any drugs.

On Day 0, your stem cells will be returned to your body by vein over 30-60 minutes.

On Days 0 through 2, you will receive palifermin by vein over about 30 seconds each day.

Beginning on Day 5, you will receive filgrastim (a drug that helps with the growth of white blood cells) through a needle under your skin 1 time each day until your blood cell levels return to normal.

Study Tests:

While you are in the hospital, you will be checked for any side effects as part of your standard of care. Blood (about 2 teaspoons) will be drawn every day to check for side effects.

As part of standard care, you will remain in the hospital for about 3-4 weeks after the transplant. After you are released from the hospital, you must remain in the Houston area to be monitored for infections and other transplant side effects until about Day 30. During this time, you will return to the clinic 1 time each week and the following tests and procedures will be performed:

* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a lung function test about 30-100 days after the transplant.

Length of Study:

You will be followed as part as the study for at least 2 years. You may be taken off study early if the disease gets worse or you experience any intolerable side effects.

At each follow-up visit the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease.
* Bone survey: Only once a year.

You must talk to the study doctor if you want to leave the study early. It may be life-threatening to leave the study after you have begun to receive the study drugs but before you receive the stem cells.

This is an investigational study. Busulfan, gemcitabine, and melphalan are all FDA approved and commercially available for the treatment of lymphoma, myeloma, and several other tumors. The use of these study drugs together and the use of gemcitabine at the dose level used in this study is investigational.

Up to 75 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years.
2. Patients with myeloma treated with first-line therapy including lenalidomide, bortezomib or thalidomide, and one or more of the following: 2.1) M paraprotein greater than 1 g/dL at HDC. 2.2) Less than partial response to first-line therapy. 2.3) Relapse after first-line therapy. 2.4) Relapse after a prior autologous stem-cell transplant.
3. Adequate renal function, as defined by serum creatinine </=1.8 mg/dL and/or estimated serum creatinine clearance >/=50 ml/min
4. Adequate hepatic function, as defined by serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) </=3 x upper limit of normal; serum bilirubin and alkaline phosphatase </=2 x upper limit of normal, unless proven to be due to disease involvement.
5. Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) >/=50% of expected corrected for hemoglobin and/or volume.
6. Adequate cardiac function with left ventricular ejection fraction >/=40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
7. Zubrod performance status <2.
8. Negative Beta human chorionic gonadotropin (HCG) text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization

Exclusion Criteria:

1. Patients with grade >/= 3 non-hematologic toxicity from previous therapy that has not resolved to </= grade 1.
2. Patients with prior whole brain irradiation
3. Patients with active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/=10,000 copies/mL, or >/= 2,000 IU/mL).
4. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
5. Active infection requiring parenteral antibiotics.
6. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal cluster of differentiation 4 (CD4) counts
7. Patients having received radiation therapy to head and neck (excluding eyes), and internal organs of chest, abdomen or pelvis in the month prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nieto Y, Valdez BC, Pingali SR, Bassett R, Delgado R, Nguyen J, Shah N, Popat U, Jones RB, Andersson BS, Gulbis A, Ahmed S, Bashir Q, Parmar S, Patel K, Myers A, Rondon G, Orlowski RZ, Champlin R, Qazilbash M. High-dose gemcitabine, busulfan, and melphalan for autologous stem-cell transplant in patients with relapsed or refractory myeloma: a phase 2 trial and matched-pair comparison with melphalan. Lancet Haematol. 2017 Jun;4(6):e283-e292. doi: 10.1016/S2352-3026(17)30080-7. Epub 2017 May 15. PMID 28522110
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the University of Texas MD Anderson Cancer Center. Out of 75, 1 participant died before starting the treatment.
Groups:
- Gemcitabine/Busulfan/Melphalan: Patients ages 18-70 with primary refractory or relapsed myeloma, candidates for an autologous SCT (ASCT) who had previously received treatment with bortezomib, an immunomodulatory drug, or both, or who were receiving a salvage ASCT.
Period: Overall Study
Arm/Group | Gemcitabine/Busulfan/Melphalan
Started | 75
Completed | 74
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine/Busulfan/Melphalan
Number analyzed (Participants) | 74
Age, Continuous [Median (Standard Deviation); unit: years] | 58.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74
Overall study group [Number; unit: participants]
  1st SCT/salvage SCT | 13
  Poor-risk cytogenetics | 6
  Extramedullary disease | 1
  Double refractory (IMiDs + proteasome inhibitors) | 11
  Disease Status: Primary refractory | 4
  Disease Status: Refractory relapse | 11
  Disease Status: Sensitive relapse | 4
  Response at ASCT: Response | 8
  Response at ASCT: Refractory | 11
  No. prior lines of treatment | 10
  No. prior lines of treatment > 2 | 9
  Post-ASCT maintenance | 16

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Had Measurable Disease at Time of Transplant and Achieved a Stringent Complete Remission
Description: Stringent complete remission was defined as negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, 5% or fewer plasma cells in bone marrow, normal free light chain ratio, and the absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Time Frame: 100 days post-transplant
Population: Only 65 participants had measurable disease at the time of ASCT.
Measure: Count of Participants; unit: Participants
Groups:
- Gemcitabine/Busulfan/Melphalan: Patients with refractory or relapsed myeloma received high-dose GemBuMel with ASCT
Arm/Group | Gemcitabine/Busulfan/Melphalan
Number analyzed (Participants) | 65
Participants | 16

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Number of participants remain free of progression or death after ASCT
Time Frame: From date of transplant until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine/Busulfan/Melphalan
Number analyzed (Participants) | 74
Participants | 31

3. Secondary Outcome: Overall Survival
Description: Number of participants from ASCT to death or last contact
Time Frame: From date of transplant until the date of death from any cause, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine/Busulfan/Melphalan
Number analyzed (Participants) | 74
Participants | 49

4. Secondary Outcome: Percent of Participants Dying From Treatment-Related Complications
Description: Participants who died from treatment-related complications from the time of ASCT.
Time Frame: From date of transplant until the date of death from treatment-related complications, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine/Busulfan/Melphalan
Number analyzed (Participants) | 74
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: All-Cause Mortality was monitored in for all enrolled 75 participants ( 1 participant died before receiving treatment and 4 while on study) and 74 participants with Serious and Other Adverse Events.
Groups:
- Gemcitabine/Busulfan/Melphalan: Participants with refractory or relapsed myeloma received high-dose GemBuMel with ASCT.
Arm/Group | Gemcitabine/Busulfan/Melphalan
All-Cause Mortality (participants affected / at risk) | 5/75
Serious Adverse Events (participants affected / at risk) | 31/74
Other Adverse Events (participants affected / at risk) | 71/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine/Busulfan/Melphalan (N=74)
Mucositis (Gastrointestinal disorders) | 13
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Diarrhea (Gastrointestinal disorders) | 2
Infection (Infections and infestations) | 5
Cardiac (Cardiac disorders) | 2
Hyperbilirubinemia (Hepatobiliary disorders) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine/Busulfan/Melphalan (N=74)
Mucositis (Gastrointestinal disorders) | 55
Dermatitis (Skin and subcutaneous tissue disorders) | 34
Diarrhea (Gastrointestinal disorders) | 13
Infection (Immune system disorders) | 71
Cardiac (Cardiac disorders) | 54
Hyperbilirubinemia (Hepatobiliary disorders) | 9
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT01237951/Prot_SAP_000.pdf